CLINICAL TRIAL: NCT04701658
Title: A Prospective Cohort Study to Evaluate the Real-world Effectiveness of Bamlanivimab in Participants With Mild-to-moderate COVID-19 at High Risk for Progressing to Severe Illness, With Matched Controls
Brief Title: A Real World Study of Bamlanivimab in Participants With Mild-to-Moderate Coronavirus Disease 2019 (COVID-19)
Acronym: BLAZE-5
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Collaborators: AbCellera Biologics Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 18216; J2X-MC-PYAJ (Other: Eli Lilly and Company)
Record Dates: First submitted 2021-01-07; First posted 2021-01-08 (Actual); Results first posted 2021-11-16 (Actual); Last update posted 2021-11-16 (Actual); Status verified 2021-11

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19 | interventions — bamlanivimab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Bamlanivimab (Experimental): Participants received 700 milligram single intravenous infusion of Bamlanivimab.
  Interventions: Drug: Bamlanivimab
- Controls (No Intervention): Matched controls who received standard of care.
  [The study was originally designed to include a matched control arm. However, due to low enrollment, it was amended to be a single arm study with Bamlanivimab arm only. No matched controls were utilized.]

INTERVENTIONS:
Drug: Bamlanivimab — Administered intravenously.
  Other Names: LY3819253; LY-CoV555
  Arms: Bamlanivimab

SUMMARY:
The purpose of this study is to find out whether bamlanivimab is able to stop COVID-19 from getting worse. Participants with mild-to-moderate COVID-19 will receive bamlanivimab via an injection into a vein. These participants will be matched to similar COVID-19 patients who received other treatment at a local medical center. All participants will be followed to learn how their disease responds. Participation could last about 3 months and includes two required visits to the study site, with the remainder of assessments performed by phone or by medical record review.

ELIGIBILITY:
Inclusion Criteria:

* Are currently not hospitalized.
* Have one or more mild or moderate COVID-19 symptoms.
* Must have first positive severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) viral infection determination and as soon as possible within 10 days of symptom onset
* Are males or non-breastfeeding females.
* Contraceptive use by males or females should be consistent with local regulations for those participating in clinical studies.
* Are at high risk for progressing to severe COVID-19 and/or hospitalization.

Exclusion Criteria:

* Participants who:

  * are hospitalized due to COVID-19, OR
  * require oxygen therapy due to COVID-19, OR
  * require an increase in baseline oxygen flow rate due to COVID-19 in those on chronic oxygen therapy due to underlying non-COVID-19 related comorbidity.
* Have peripheral capillary oxygen saturation (SpO2) less than or equal to (≤) 90 percent on room air or arterial partial pressure of oxygen/fraction of inspired oxygen (PaO2/FiO2) less than (<) 300, respiratory rate greater than or equal to (≥) 30 per minute, heart rate ≥125 per minute.
* Have body weight <40 kilograms.
* Require mechanical ventilation or anticipated impending need for mechanical ventilation.
* Have known allergies to any of the components used in the formulation of the interventions.
* Suspected or proven serious, active bacterial, fungal, viral, or other infection (besides COVID-19) that in the opinion of the investigator could constitute a risk when taking intervention.
* Have any comorbidity requiring surgery within <7 days, or that is considered life-threatening within 29 days.
* Have any serious concomitant systemic disease, condition, or disorder that, in the opinion of the investigator, should preclude participation in this study.
* Have a history of a positive SARS-CoV-2 serology test.
* Have a history of a positive SARS-CoV-2 test prior to the one serving as eligibility for this study.
* Have received an investigational intervention for SARS-CoV-2 prophylaxis within 30 days before dosing.
* Have received treatment with a SARS-CoV-2-specific monoclonal antibody, remdesivir, or other treatment for COVID-19.
* Have received convalescent COVID-19 plasma treatment.
* Have participated in a previous SARS-CoV-2 vaccine study.
* Have participated, within the last 30 days, in a clinical study involving an investigational intervention. If the previous investigational intervention has a long half-life, 5 half-lives or 30 days, whichever is longer, should have passed.
* Are concurrently enrolled in any other type of medical research judged not to be scientifically or medically compatible with this study.
* Are breast-feeding.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 109 (Actual)
Dates: Start 2021-02-01 (Actual); Primary Completion 2021-06-22 (Actual); Study Completion 2021-06-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- Presbyterian Medical Center, Albuquerque, New Mexico, United States

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual patient level data will be provided in a secure access environment upon approval of a research proposal and a signed data sharing agreement.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data are available 6 months after the primary publication and approval of the indication studied in the US and European Union (EU), whichever is later. Data will be indefinitely available for requesting.
Access Criteria: A research proposal must be approved by an independent review panel and researchers must sign a data sharing agreement.
URL: http://vivli.org/

REFERENCES:
- [Derived] Kreuzberger N, Hirsch C, Chai KL, Tomlinson E, Khosravi Z, Popp M, Neidhardt M, Piechotta V, Salomon S, Valk SJ, Monsef I, Schmaderer C, Wood EM, So-Osman C, Roberts DJ, McQuilten Z, Estcourt LJ, Skoetz N. SARS-CoV-2-neutralising monoclonal antibodies for treatment of COVID-19. Cochrane Database Syst Rev. 2021 Sep 2;9(9):CD013825. doi: 10.1002/14651858.CD013825.pub2. PMID 34473343
- See also: A Real World Study of Bamlanivimab in Participants With Mild-to-moderate Coronavirus Disease 2019 (COVID-19) (BLAZE-5) — https://trials.lillytrialguide.com/en-US/trial/7zjYxdhUwux6y1A18CmrFJ

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was originally designed to include a matched control arm. However, due to low enrollment, it was amended to be a single arm study with Bamlanivimab arm only. No matched controls were utilized.
Groups:
- Bamlanivimab 700 Milligram (mg): Participants received 700 mg single intravenous (IV) infusion of Bamlanivimab.
Period: Overall Study
Arm/Group | Bamlanivimab 700 Milligram (mg)
Started | 109
Received Single Dose of Bamlanivimab | 109
Completed | 103
Not Completed | 6
Not completed — Lost to Follow-up | 6

BASELINE CHARACTERISTICS:
Population: All participants who received single dose of Bamlanivimab.
Groups:
- Bamlanivimab 700 mg: Participants received 700 mg single IV infusion of Bamlanivimab.
Arm/Group | Bamlanivimab 700 mg
Number analyzed (Participants) | 109
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.40 (15.34)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 61
  Male | 48
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 50
  Not Hispanic or Latino | 55
  Unknown or Not Reported | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 3
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 1
  Black or African American | 6
  White | 83
  More than one race | 1
  Unknown or Not Reported | 13
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 109

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Who Experience COVID-19 Related Hospitalization or Death From Any Cause
Description: Percentage of Participants who Experience COVID-19 Related Hospitalization or Death From Any Cause. Hospitalization is defined as ≥24 hours of acute care.
Time Frame: Baseline through Days 29, 60, and 90
Population: All participants who received single dose of Bamlanivimab.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Bamlanivimab 700 mg
Number analyzed (Participants) | 109
Percentage of participants
  Baseline through Day 29 | 0.9 [0 to 2.7]
  Baseline through Day 60 | 0.9 [0 to 2.7]
  Baseline through Day 90 | 0.9 [0 to 2.7]

2. Secondary Outcome: Percentage of Participants With a COVID-19-related Hospitalization
Description: Hospitalization is defined as ≥24 hours of acute care.
Time Frame: Baseline through Days 29, 60, and 90
Population: All participants who received single dose of Bamlanivimab.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Bamlanivimab 700 mg
Number analyzed (Participants) | 109
Percentage of participants
  Baseline through Day 29 | 0.9 [0 to 2.7]
  Baseline through Day 60 | 0.9 [0 to 2.7]
  Baseline through Day 90 | 0.9 [0 to 2.7]

3. Secondary Outcome: Percentage of Participants With a COVID-related Emergency Department (ED) Visit
Description: Percentage of Participants with a COVID-related ED Visit.
Time Frame: Baseline through Days 29, 60, and 90
Population: All participants who received single dose of Bamlanivimab.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Bamlanivimab 700 mg
Number analyzed (Participants) | 109
Percentage of participants
  Baseline through Day 29 | 5.5 [1.2 to 9.8]
  Baseline through Day 60 | 5.5 [1.2 to 9.8]
  Baseline through Day 90 | 5.5 [1.2 to 9.8]

ADVERSE EVENTS:
Time Frame: Baseline through Follow-up (Up to 90 days)
Description: All participants who received single dose of Bamlanivimab.
Arm/Group | Bamlanivimab 700 mg
All-Cause Mortality (participants affected / at risk) | 0/109
Serious Adverse Events (participants affected / at risk) | 2/109
Other Adverse Events (participants affected / at risk) | 9/109
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Bamlanivimab 700 mg (N=109)
Cholelithiasis (Hepatobiliary disorders) | 1 (1)
End stage renal disease (Renal and urinary disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Bamlanivimab 700 mg (N=109)
Tachycardia (Cardiac disorders) | 1 (1)
Vision blurred (Eye disorders) | 1 (1)
Infusion site extravasation (General disorders) | 5 (5)
Headache (Nervous system disorders) | 1 (1)
Paranasal sinus hypersecretion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pharyngeal swelling (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
The study was originally designed to include a matched control arm. However, due to low enrollment, it was amended to be a single arm study with Bamlanivimab arm only. No matched controls were utilized. Therefore, no comparative analyses were conducted. All analyses were descriptive in nature and conducted only on Bamlanivimab-treated participants.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2020-12-18): https://cdn.clinicaltrials.gov/large-docs/58/NCT04701658/Prot_000.pdf
  • Statistical Analysis Plan (2021-08-13): https://cdn.clinicaltrials.gov/large-docs/58/NCT04701658/SAP_001.pdf